CLINICAL TRIAL: NCT04124874
Title: Prevalence and Impact on Quality of Life of Lower Urinary Tract Symptoms (LUTS) in Night Workers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jagiellonian University (Other)
Collaborators: Piotr Chlosta (Unknown)
Responsible Party: Principal Investigator, Mikolaj Przydacz, Assistant, Jagiellonian University
Other Study IDs: 1072.6120.200.2019
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: To Evaluate Lower Urinary Tract Symptoms (LUTS) and Their Impact on Quality of Life in Night Workers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There will be no intervention — There will be no intervention

SUMMARY:
The first large population-based study to evaluate lower urinary tract symptoms and their impact on quality of life in night workers.

DETAILED DESCRIPTION:
The first large population-based study to evaluate lower urinary tract symptoms (LUTS) and their impact on quality of life in night workers. The study objective is to assess the prevalence and bother of LUTS in the population of night workers.

This study will be conducted as a questionnaire survey with assessment of LUTS using a standardized protocol based on definitions by the International Continence Society (ICS). The International Prostate Symptom Score (IPSS), the Overactive Bladder- Validated 8-question Screener (OAB-V8), the Patient Health Questionnaire-9 (PHQ-9), the Athen Insomnia Scale, the Work Productivity and Activity Impairment Questionnaire (WPAI), the 12-Item Short Form Health Survey (SF-12) questionnaires will be included. Participants will be also asked to rate how often they experienced individual LUTS and the degree of associated bother.

ELIGIBILITY:
Inclusion Criteria:

Night workers defined as any workers, who, during night time, work at least three hours of their daily working time as a normal course or who work at night at least 1/4 of their working time during the accounting period (definition by the Polish Labour Code).

Exclusion Criteria:

Non night workers Urinary tract infection in the past 4 weeks

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Night workers defined as any workers, who, during night time, work at least three hours of their daily working time as a normal course or who work at night at least 1/4 of their working time during the accounting period (definition by the Polish Labour Code).
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of LUTS | Through study completion, an average of 3 months
  The prevalence of LUTS will be assessed using definitions of the International Continence Society (descriptive statistics).
Symptom bother of LUTS | Through study completion, an average of 3 months
  The degree of associated bother will be assessed using Likert scale (Likert scale: not at all [score 0], a little bit [score 1], somewhat [score 2], quite a bit [score 3], a great deal [score 4], or a very great deal [score 5]).

SECONDARY OUTCOMES:
Prevalence of specific lower urinary tract symptoms | Through study completion, an average of 3 months
  The prevalence of specific lower urinary tract symptoms will be assessed using a standardised protocol based on the definitions provided by the International Continence Society (i.e. storage symptoms, voiding symptoms and post-micturition symptoms).
Symptom bother of specific lower urinary tract symptoms | Through study completion, an average of 3 months
  The degree of associated bother of specific lower urinary tract symptoms will be assessed using Likert scale (Likert scale: not at all [score 0], a little bit [score 1], somewhat [score 2], quite a bit [score 3], a great deal [score 4], or a very great deal [score 5]).
Prevalence of OAB | Through study completion, an average of 3 months
  The prevalence of OAB will be assessed with the Overactive Bladder-Validated 8-question Screener (OAB- V8) questionnaire.
Prevalence of depressive symptoms | Through study completion, an average of 3 months
  The prevalence of depressive symptoms will be assessed with the PHQ-9 (Patient Health Questionnaire-9).
Sleep quality | Through study completion, an average of 3 months
  The sleep quality will be assessed with the Athen Insomnia Scale questionnaire.
Work productivity | Through study completion, an average of 3 months
  The work productivity will be assessed with the Work Productivity and Activity Impairment Questionnaire (WPAI).
General quality of life | Through study completion, an average of 3 months
  The general quality of life will be assessed with the 12-Item Short Form Health Survey (SF-12).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology Jagiellonian University, Krakow, Poland